CLINICAL TRIAL: NCT01737099
Title: Efficacy and Safety Study of DHA-O in Adults With Hypertriglyceridemia
Acronym: DHA-O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-1048
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Hypertriglyceridemia
Keywords: omega-3; DHA; triglycerides; lipids; cardiovascular; hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DHA-O (Experimental)
  Interventions: Dietary Supplement: DHA-O
- Fish oil (Active Comparator)
  Interventions: Dietary Supplement: Fish oil
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DHA-O
  Arms: DHA-O
Dietary Supplement: Fish oil
  Arms: Fish oil
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of DHA-O to lower elevated triglyceride levels in healthy adults with hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-79
* fasting TG levels, 150-499 mg/dL
* baseline DHA intake <200mg/d
* active and in good health

Exclusion Criteria:

* recent diagnosis of CHD or history of revascularization within 6mos of study
* use of lipid altering medications (other than stable statins)
* use of anticoagulants
* use of omega-3 products within 4 weeks of screening
* serum AST/ALT >1.5x ULN and/or creatinine >1.5 mg/dL at screening
* lipid altering foods or supplements
* women who are pregnant or of childbearing potential not using adequate birth control
* current use or history of drug or alcohol abuse
* inability to swallow capsules

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in TG levels | week 14

SECONDARY OUTCOMES:
Change from baseline in lipid panel measures | week 14

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Principal Investigator — Biofortis Clinical Research, Inc.
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

REFERENCES:
- [Derived] Maki KC, Yurko-Mauro K, Dicklin MR, Schild AL, Geohas JG. A new, microalgal DHA- and EPA-containing oil lowers triacylglycerols in adults with mild-to-moderate hypertriglyceridemia. Prostaglandins Leukot Essent Fatty Acids. 2014 Oct;91(4):141-8. doi: 10.1016/j.plefa.2014.07.012. Epub 2014 Jul 22. PMID 25123060